CLINICAL TRIAL: NCT05410288
Title: A Clinical Investigation of the Effects of Acu-TENS and Acupressure on the Sleep Quality of Older Adults With Insomnia: A Pilot Randomized, Placebo-controlled Clinical Trial
Brief Title: Acu-TENS and Acupressure on the Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Assoc. Head(RS), ADoRCMI & Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022ShamayAcu-tens
Record Dates: First submitted 2022-05-31; First posted 2022-06-08 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: acuTENS; Sleep Quality; Insomnia; Acupressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain assessor blinding, all interventions will be delivered by the part-time research assistant with health-related education background. All assessments and data entry will be performed by an independent full-time research assistant. In addition, the treatment and assessment will be conducted at different sites. Any analysts or statisticians involved in data management will also be blinded to the identification of each treatment group until the final efficacy analysis for each treatment group has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acu-TENS+SHP (Experimental): Participants in the Acu-TENS group will receive Acu-TENS coupled with a sleep hygiene program (SHP). 4 weeks and comprise thrice-weekly 30-min sessions.
  Interventions: Device: Acu-TENS; Other: sleep hygiene program(SHP)
- acupressure+SHP (Experimental): The acupressure group will receive acupressure and SHP. 4 weeks and comprise thrice-weekly 30-min sessions.
  Interventions: Other: acupressure+SHP; Other: sleep hygiene program(SHP)
- placebo stimulation+SHP (Placebo Comparator): The placebo group will receive a placebo stimulation and SHP. 4 weeks and comprise thrice-weekly 30-min sessions.
  Interventions: Other: placebo stimulation+SHP; Other: sleep hygiene program(SHP)

INTERVENTIONS:
Device: Acu-TENS — A TENS stimulator will be used (NeuroTrac TENS; Verity Medical Ltd., Wexford, Ireland). Electrodes will be placed over selected acupoints (i.e., bilateral SP6, PC6 and HT7) and connected to the TENS stimulator. These acupoints are selected according to the traditional Chinese medicine and results of previous studies. The stimulation will be lasted 30-min for each session. The frequency of the stimulation parameter's waveform will be set to 100 Hz and the square pulses will be set to 0.2-ms. The intensity of the stimulation will be below motor threshold and lower than the intolerable level, and hence, participants will feel a pleasant and mild aching sensation.
  Arms: Acu-TENS+SHP
Other: acupressure+SHP — Participants in the acupressure group will receive acupressure coupled with SHP. The acupressure protocol was developed based on a protocol recommended by a review and will comprise the following: (1) applying consistent finger-tip pressure of 3-5 kg, with rotational movements; (2) counterclockwise and then clockwise circular motions for 2.5-min each; (3) confirming the precision of the acupressure based on participants feeling pain, numbness, distension, or warmth at the point of application; and (4) an acupoint sequence from the leg to the head, first on the left side of the body and then on the right side of the body; and (5) a 5-min treatment on each acupoint (i.e., bilateral SP6, PC6, and HT7) in each 30-min session. The SHP is the same with Acu-TENS+SHP group.
  Arms: acupressure+SHP
Other: placebo stimulation+SHP — Participants in the placebo stimulation + SHP group will receive 30-minute placebo stimulation from identical-looking TENS devices with the electrical circuit disconnected inside.
  Arms: placebo stimulation+SHP
Other: sleep hygiene program(SHP) — SHP is a set of instructions designed to help with sleep and promote healthy sleeping habits. The sleep guide contains information on how much sleep is needed by every individual daily, factors that could affect sleep, and risk factors for sleep disorders. It also contains information on the types of sleep disorders, delayed sleep syndrome, insomnia-producing behavior that could affect sleep quality, and suggestions for inducing sleep. The participants will be instructed to read the guide after the baseline assessment (T0). Those instructions will be reinforced by the research practitioner after each treatment session, in order to maintain the healthy sleeping habits.

SUMMARY:
The study aims to investigate the effects of two non-invasive acupuncture methodologies applied to three selected acupoints on the sleep quality of older adults with insomnia.

The investigators invite participants to participate in the study (12 treatments [3 times/week, 4 weeks in total], 3 tests), which will take about 2 months in total. Participants will be randomly allocated to three independent groups, i.e., a placebo group or one of two treatment groups, viz., a transcutaneous electrical nerve-stimulation group (Acu-TENS) or an acupressure group. The Acu-TENS group will receive Acu-TENS + a sleep hygiene program (SHP). The acupressure group will receive acupressure + SHP. The placebo group will receive a placebo stimulation+ SHP. Each group will have a 4-week treatment comprising thrice-weekly 30-min sessions of treatment.

For Acu-TENS, electrodes will be attached to participants' sleep-related acupoints for 30 minutes. For acupressure, the investigators will guide participants to apply pressure to each sleep-related acupoint for 5 minutes, for a total of 30 minutes. The process of Sham Acu-TENS stimulation will be the same as Acu-TENS, but the instrument model is different. SHP is a training course in which the investigators will guide participants on how to improve participants' sleep quality by adjusting participants' lifestyle. The sleep quality (survey and actigraphy), insomnia index, heart rate variability, level of fatigue (survey), mood (survey) and quality of life (survey) will be measured at the baseline assessment (before the treatment), post-treatment assessment (after the four weeks treatment) and follow-up assessment (two weeks after the treatment ended). The investigators will give participants a watch to wear for one week during sleep measurement and then please return it. The watch will record participants' sleep data. For the heart rate variability measurement, participants will need to wear a heart rate monitor in the lab for a short period. After the trials, Participants will have the opportunity to know participants' level of sleep quality and some mental conditions (i.e., mood, fatigue, quality of life). Participants may experience mild skin irritation during treatment. If participants feel uncomfortable, please inform the researcher to reduce the irritation to a relatively comfortable level.

DETAILED DESCRIPTION:
Insomnia is the most common sleep disorder that affects older adults. This proposed study aims to investigate the effects of two acupuncture methodology applied to three selected acupoints on the sleep quality of older adults with insomnia. The study will be a single-blind randomized controlled trial with a pre-post design and involve three parallel groups of older adult participants (aged > 55 years) diagnosed with insomnia. The participants will be randomly allocated to three independent groups, i.e., a placebo group or one of two treatment groups, viz., a transcutaneous electrical nerve-stimulation group (Acu-TENS) or an acupressure group. The Acu-TENS group will receive a 4-week treatment comprising thrice-weekly 30-min sessions of Acu-TENS + a sleep hygiene program (SHP). The acupressure group will receive acupressure + SHP. The selected acupoints will be bilateral Sanyinjiao (SP6) on the legs and Shenmen (HT7) and Neiguan (PC6) on the wrists. The placebo group will receive a placebo stimulation+ SHP. The primary outcomes of the study will be sleep quality, insomnia index as well as actigraphy. The secondary outcomes will be heart rate variability, level of fatigue, mood, and quality of life. All the outcomes will be measured at the baseline assessment (before the treatment), post-treatment assessment (after the four weeks treatment) and follow-up assessment (two weeks after the treatment ended). It is hypothesized that the Acu-TENS + SHP treatment will better alleviate insomnia in participants than acupressure + SHP or placebo stimulation + SHP.

ELIGIBILITY:
Inclusion Criteria:

* aged 55 years or older; and
* self-reported poor sleep quality (PSQI, scores ≥ 6) in the past 4 weeks

Exclusion Criteria:

* an amputation or recent fracture of upper or lower limbs;
* a severe disease that precludes the receipt of Acu-TENS or acupressure (e.g., renal impairment; epilepsy; cardiac pace-mark or another electrical or metal implant in participants' body);
* taking medication that may affect sleep;
* skin lesions, infection, or inflammation near selected acupoints; or
* a psychiatrically diagnosed mental disease.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | T0, baseline
  The Pittsburgh sleep quality index is a 19-item self-report survey designed to assess subjective sleep quality across 4 weeks. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Pittsburgh sleep quality index (PSQI) | T1, post (4th week)
  The Pittsburgh sleep quality index is a 19-item self-report survey designed to assess subjective sleep quality across 4 weeks. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Pittsburgh sleep quality index (PSQI) | T2, follow-up(6th week)
  The Pittsburgh sleep quality index is a 19-item self-report survey designed to assess subjective sleep quality across 4 weeks. It has been used in both research and clinical settings to evaluate sleep quality and screen for sleep disturbances. The scores ranges from 0 to 21. A higher score means a lower sleep quality, with a score ≥ 6 as the cut-off value for poor sleep quality. The Chinese version will be used in the proposed study.
Insomnia severity index (ISI) | T0, baseline
  The ISI is a self-report survey designed to assess the subjective perception of the severity of insomnia. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.
Insomnia severity index (ISI) | T1, post (4th week)
  The ISI is a self-report survey designed to assess the subjective perception of the severity of insomnia. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.
Insomnia severity index (ISI) | T2, follow-up(6th week)
  The ISI is a self-report survey designed to assess the subjective perception of the severity of insomnia. It comprises seven items measuring the severity of sleep-onset and sleep maintenance difficulties (both nocturnal and early-morning awakenings), satisfaction with the current sleep pattern, the adverse effects of insomnia on daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a scale from 0 to 4, and the total score ranges from 0 to 28. A higher score represents more severe insomnia. The Chinese version will be used in the proposed study.
Total sleep time | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' total sleep time (total time asleep from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Total sleep time | T1, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' total sleep time (total time asleep from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Total sleep time | T2, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' total sleep time (total time asleep from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Sleep efficiency | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' sleep efficiency (percentage of total time in bed trying to sleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Sleep efficiency | T1, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' sleep efficiency (percentage of total time in bed trying to sleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Sleep efficiency | T2, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants' sleep efficiency (percentage of total time in bed trying to sleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Sleep onset latency | T1, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'sleep onset latency (time to fall asleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Sleep onset latency | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'sleep onset latency (time to fall asleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Sleep onset latency | T2, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'sleep onset latency (time to fall asleep). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Time awake after sleep onset | T1, post (4th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'time awake after sleep onset (total time awake from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Time awake after sleep onset | T0, baseline
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'time awake after sleep onset (total time awake from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.
Time awake after sleep onset | T2, follow-up(6th week)
  Actigraphy (Ambulatory Monitoring, Inc., Ardsley, NY, or equivalent device) will be used to measure participants'time awake after sleep onset (total time awake from sleep onset to waking). Actigraphy is a non-invasive technique that involves the use of a wearable device to objectively measure sleep in terms of ambulation. Thus, actigraphic sleep metrics are based on the principle that sleep is characterized by the relative absence of movement. Participants will be instructed to wear an actigraphy device on one of their legs and press the event-marker to record bedtimes and rise time for three consecutive days at each assessment point (i.e., T0, T1, T2). The validity of this assessment was confirmed in previous research.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | T0, baseline
  Heart rate and heart rate variability will be measured by electrocardiography (ECG; SphygmoCor, AtCor Medical, Sydney, Australia, or equivalent device), using a device that acquires, stores, and processes electrocardiogram signals. Participants will be measured in the morning between 8:00 to 11:00 am. The sympathetic nervous activity, and the high frequency will be used to indicate parasympathetic nervous activity.
Heart Rate Variability (HRV) | T1, post (4th week)
  Heart rate and heart rate variability will be measured by electrocardiography (ECG; SphygmoCor, AtCor Medical, Sydney, Australia, or equivalent device), using a device that acquires, stores, and processes electrocardiogram signals. Participants will be measured in the morning between 8:00 to 11:00 am. The sympathetic nervous activity, and the high frequency will be used to indicate parasympathetic nervous activity.
Heart Rate Variability (HRV) | T2, follow-up(6th week)
  Heart rate and heart rate variability will be measured by electrocardiography (ECG; SphygmoCor, AtCor Medical, Sydney, Australia, or equivalent device), using a device that acquires, stores, and processes electrocardiogram signals. Participants will be measured in the morning between 8:00 to 11:00 am. The sympathetic nervous activity, and the high frequency will be used to indicate parasympathetic nervous activity.
Depression Anxiety Stress Scale | T0, baseline
  Participants' mood will be measured using the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
Depression Anxiety Stress Scale | T1, post (4th week)
  Participants' mood will be measured using the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
Depression Anxiety Stress Scale | T2, follow-up(6th week)
  Participants' mood will be measured using the Depression Anxiety Stress Scale, a 21-item survey that assesses depression, anxiety, and stress. Each index (i.e., depression, anxiety, and stress) comprises seven items. The scores ranges from 0 to 42. Higher score indicates more sever symptom. The reliability of this scale was confirmed in previous research.
The Fatigue Assessment Scale | T0, baseline
  The Fatigue Assessment Scale will be used to measure participants' general fatigue. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
The Fatigue Assessment Scale | T1, post (4th week)
  The Fatigue Assessment Scale will be used to measure participants' general fatigue. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
The Fatigue Assessment Scale | T2, follow-up(6th week)
  The Fatigue Assessment Scale will be used to measure participants' general fatigue. It is a 10-item survey, of which 5 items assess physical fatigue and the remaining 5 items assess mental fatigue. The total score ranges from 10 to 50, and a total score ≥ 22 indicates fatigue. The translated Chinese version will be used in the proposed study.
Health-related Quality of Life (QoL) | T0, baseline
  The 12-item Short-Form Survey will be used to measure participants' QoL. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL. The translated Cantonese version will be used in this proposed study .
Health-related Quality of Life (QoL) | T1, post (4th week)
  The 12-item Short-Form Survey will be used to measure participants' QoL. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL. The translated Cantonese version will be used in this proposed study .
Health-related Quality of Life (QoL) | T2, follow-up(6th week)
  The 12-item Short-Form Survey will be used to measure participants' QoL. This instrument contains eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The total score ranges from 0 to 100, with a higher score indicating better QoL. The translated Cantonese version will be used in this proposed study .

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao H, Pan X, Li H, Liu J. Acupuncture for treatment of insomnia: a systematic review of randomized controlled trials. J Altern Complement Med. 2009 Nov;15(11):1171-86. doi: 10.1089/acm.2009.0041. PMID 19922248
- [Background] Chiou YF, Yeh ML, Wang YJ. Transcutaneous Electrical Nerve Stimulation on Acupuncture Points Improves Myofascial Pain, Moods, and Sleep Quality. Rehabil Nurs. 2020 Jul/Aug;45(4):225-233. doi: 10.1097/RNJ.0000000000000198. PMID 30694996
- [Background] Crowley K. Sleep and sleep disorders in older adults. Neuropsychol Rev. 2011 Mar;21(1):41-53. doi: 10.1007/s11065-010-9154-6. Epub 2011 Jan 12. PMID 21225347
- [Background] Flachskampf FA, Gallasch J, Gefeller O, Gan J, Mao J, Pfahlberg AB, Wortmann A, Klinghammer L, Pflederer W, Daniel WG. Randomized trial of acupuncture to lower blood pressure. Circulation. 2007 Jun 19;115(24):3121-9. doi: 10.1161/CIRCULATIONAHA.106.661140. Epub 2007 Jun 4. PMID 17548730
- [Background] Fu CW, Shu Q, Jiao Y, Wu T, Song AQ, Zhu QC, Zhang WP. A comparison of noninvasive and invasive acupuncture in preventing postoperative nausea and vomiting: A protocol for systematic review and Bayesian network meta-analysis. Medicine (Baltimore). 2020 Jul 31;99(31):e21544. doi: 10.1097/MD.0000000000021544. PMID 32756210
- [Background] Gibson W, Wand BM, Meads C, Catley MJ, O'Connell NE. Transcutaneous electrical nerve stimulation (TENS) for chronic pain - an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2019 Feb 19;2(2):CD011890. doi: 10.1002/14651858.CD011890.pub2. PMID 30776855
- [Background] He W, Li M, Zuo L, Wang M, Jiang L, Shan H, Han X, Yang K, Han X. Acupuncture for treatment of insomnia: An overview of systematic reviews. Complement Ther Med. 2019 Feb;42:407-416. doi: 10.1016/j.ctim.2018.12.020. Epub 2018 Dec 28. PMID 30670275
- [Background] He Y, Guo X, May BH, Zhang AL, Liu Y, Lu C, Mao JJ, Xue CC, Zhang H. Clinical Evidence for Association of Acupuncture and Acupressure With Improved Cancer Pain: A Systematic Review and Meta-Analysis. JAMA Oncol. 2020 Feb 1;6(2):271-278. doi: 10.1001/jamaoncol.2019.5233. PMID 31855257
- [Background] Johnson MI, Bjordal JM. Transcutaneous electrical nerve stimulation for the management of painful conditions: focus on neuropathic pain. Expert Rev Neurother. 2011 May;11(5):735-53. doi: 10.1586/ern.11.48. PMID 21539490
- [Background] Kathol RG, Arnedt JT. Cognitive Behavioral Therapy for Chronic Insomnia: Confronting the Challenges to Implementation. Ann Intern Med. 2016 Jul 19;165(2):149-50. doi: 10.7326/M16-0359. Epub 2016 May 3. No abstract available. PMID 27136604
- [Background] Khan MS, Aouad R. The Effects of Insomnia and Sleep Loss on Cardiovascular Disease. Sleep Med Clin. 2017 Jun;12(2):167-177. doi: 10.1016/j.jsmc.2017.01.005. Epub 2017 Mar 25. PMID 28477772
- [Background] Kuppermann M, Lubeck DP, Mazonson PD, Patrick DL, Stewart AL, Buesching DP, Fifer SK. Sleep problems and their correlates in a working population. J Gen Intern Med. 1995 Jan;10(1):25-32. doi: 10.1007/BF02599573. PMID 7699483
- [Background] Liu Y, Zhang J, Lam SP, Yu MW, Li SX, Zhou J, Chan JW, Chan NY, Li AM, Wing YK. Help-seeking behaviors for insomnia in Hong Kong Chinese: a community-based study. Sleep Med. 2016 May;21:106-13. doi: 10.1016/j.sleep.2016.01.006. Epub 2016 Feb 12. PMID 27448480
- [Background] Lu MJ, Lin ST, Chen KM, Tsang HY, Su SF. Acupressure improves sleep quality of psychogeriatric inpatients. Nurs Res. 2013 Mar-Apr;62(2):130-7. doi: 10.1097/NNR.0b013e3182781524. PMID 23302821
- [Background] Matthews EE, Arnedt JT, McCarthy MS, Cuddihy LJ, Aloia MS. Adherence to cognitive behavioral therapy for insomnia: a systematic review. Sleep Med Rev. 2013 Dec;17(6):453-64. doi: 10.1016/j.smrv.2013.01.001. Epub 2013 Apr 17. PMID 23602124
- [Background] Meng L, Zheng Y, Hui R. The relationship of sleep duration and insomnia to risk of hypertension incidence: a meta-analysis of prospective cohort studies. Hypertens Res. 2013 Nov;36(11):985-95. doi: 10.1038/hr.2013.70. Epub 2013 Sep 5. PMID 24005775
- [Background] Ng SS, Hui-Chan CW. Transcutaneous electrical nerve stimulation combined with task-related training improves lower limb functions in subjects with chronic stroke. Stroke. 2007 Nov;38(11):2953-9. doi: 10.1161/STROKEAHA.107.490318. Epub 2007 Sep 27. PMID 17901383
- [Background] Park JE, Lee SS, Lee MS, Choi SM, Ernst E. Adverse events of moxibustion: a systematic review. Complement Ther Med. 2010 Oct;18(5):215-23. doi: 10.1016/j.ctim.2010.07.001. Epub 2010 Aug 19. PMID 21056845
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- [Background] QuickStats: Percentage* of Adults Aged >/=18 Years Who Took Medication To Help Fall or Stay Asleep Four or More Times in the Past Week,dagger by Sex and Age Group - National Health Interview Survey, United States, 2017-2018 section sign. MMWR Morb Mortal Wkly Rep. 2019 Dec 13;68(49):1150. doi: 10.15585/mmwr.mm6849a5. No abstract available. PMID 31830011
- [Background] Siu PM, Yu AP, Tam BT, Chin EC, Yu DS, Chung KF, Hui SS, Woo J, Fong DY, Lee PH, Wei GX, Irwin MR. Effects of Tai Chi or Exercise on Sleep in Older Adults With Insomnia: A Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2037199. doi: 10.1001/jamanetworkopen.2020.37199. PMID 33587135
- [Background] Sokunbi G, Takai IU, Nwosu IB, Balarabe R. Effects of Acupressure and Acupuncture-Like Transcutaneous Electrical Nerve Stimulation on Sleep Quality Among Pregnant Women. J Acupunct Meridian Stud. 2020 Dec;13(6):180-186. doi: 10.1016/j.jams.2020.10.003. Epub 2020 Nov 1. PMID 33137517
- [Background] Sun JL, Sung MS, Huang MY, Cheng GC, Lin CC. Effectiveness of acupressure for residents of long-term care facilities with insomnia: a randomized controlled trial. Int J Nurs Stud. 2010 Jul;47(7):798-805. doi: 10.1016/j.ijnurstu.2009.12.003. Epub 2010 Jan 6. PMID 20056221
- [Background] Sun YJ, Yuan JM, Yang ZM. Effectiveness and safety of moxibustion for primary insomnia: a systematic review and meta-analysis. BMC Complement Altern Med. 2016 Jul 13;16:217. doi: 10.1186/s12906-016-1179-9. PMID 27411310
- [Background] Tao H, Wang T, Dong X, Guo Q, Xu H, Wan Q. Effectiveness of transcutaneous electrical nerve stimulation for the treatment of migraine: a meta-analysis of randomized controlled trials. J Headache Pain. 2018 May 29;19(1):42. doi: 10.1186/s10194-018-0868-9. PMID 29845369
- [Background] Tsay SL, Chen ML. Acupressure and quality of sleep in patients with end-stage renal disease--a randomized controlled trial. Int J Nurs Stud. 2003 Jan;40(1):1-7. doi: 10.1016/s0020-7489(02)00019-6. PMID 12550145
- [Background] Waits A, Tang YR, Cheng HM, Tai CJ, Chien LY. Acupressure effect on sleep quality: A systematic review and meta-analysis. Sleep Med Rev. 2018 Feb;37:24-34. doi: 10.1016/j.smrv.2016.12.004. Epub 2016 Dec 22. PMID 28089414
- [Background] Wang F, Eun-Kyoung Lee O, Feng F, Vitiello MV, Wang W, Benson H, Fricchione GL, Denninger JW. The effect of meditative movement on sleep quality: A systematic review. Sleep Med Rev. 2016 Dec;30:43-52. doi: 10.1016/j.smrv.2015.12.001. Epub 2015 Dec 12. PMID 26802824
- [Background] Wang X, Li P, Pan C, Dai L, Wu Y, Deng Y. The Effect of Mind-Body Therapies on Insomnia: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Feb 13;2019:9359807. doi: 10.1155/2019/9359807. eCollection 2019. PMID 30894878
- [Background] Wong WS, Fielding R. Prevalence of insomnia among Chinese adults in Hong Kong: a population-based study. J Sleep Res. 2011 Mar;20(1 Pt 1):117-26. doi: 10.1111/j.1365-2869.2010.00822.x. PMID 20408932
- [Background] Xu H, Shi Y, Xiao Y, Liu P, Wu S, Pang P, Deng L, Chen X. Efficacy Comparison of Different Acupuncture Treatments for Primary Insomnia: A Bayesian Analysis. Evid Based Complement Alternat Med. 2019 Sep 3;2019:8961748. doi: 10.1155/2019/8961748. eCollection 2019. PMID 31565065
- [Background] Yeung WF, Chung KF, Yung KP, Ho FY, Ho LM, Yu YM, Kwok CW. The use of conventional and complementary therapies for insomnia among Hong Kong Chinese: a telephone survey. Complement Ther Med. 2014 Oct;22(5):894-902. doi: 10.1016/j.ctim.2014.08.001. Epub 2014 Aug 8. PMID 25440381
- [Result] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Clark LA, Watson D. Tripartite model of anxiety and depression: psychometric evidence and taxonomic implications. J Abnorm Psychol. 1991 Aug;100(3):316-36. doi: 10.1037//0021-843x.100.3.316. PMID 1918611
- [Result] Hmwe NTT, Browne G, Mollart L, Allanson V, Chan SW. Acupressure to improve sleep quality of older people in residential aged care: a randomised controlled trial protocol. Trials. 2020 Apr 25;21(1):360. doi: 10.1186/s13063-020-04286-2. PMID 32334620
- [Result] Ho LYW, Lai CKY, Ng SSM. Measuring fatigue following stroke: the Chinese version of the Fatigue Assessment Scale. Disabil Rehabil. 2021 Nov;43(22):3234-3241. doi: 10.1080/09638288.2020.1730455. Epub 2020 Mar 6. PMID 32142618
- [Result] Lam ET, Lam CL, Fong DY, Huang WW. Is the SF-12 version 2 Health Survey a valid and equivalent substitute for the SF-36 version 2 Health Survey for the Chinese? J Eval Clin Pract. 2013 Feb;19(1):200-8. doi: 10.1111/j.1365-2753.2011.01800.x. Epub 2011 Nov 29. PMID 22128754
- [Result] Leger D, Guilleminault C, Bader G, Levy E, Paillard M. Medical and socio-professional impact of insomnia. Sleep. 2002 Sep 15;25(6):625-9. PMID 12224841
- [Result] Li W, Li Z, Zhang H, Wang Y, Chen H, Xiong L. Acupoint Catgut Embedding for Insomnia: A Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2020 Nov 6;2020:5450824. doi: 10.1155/2020/5450824. eCollection 2020. PMID 33204287
- [Result] Ohayon M, Wickwire EM, Hirshkowitz M, Albert SM, Avidan A, Daly FJ, Dauvilliers Y, Ferri R, Fung C, Gozal D, Hazen N, Krystal A, Lichstein K, Mallampalli M, Plazzi G, Rawding R, Scheer FA, Somers V, Vitiello MV. National Sleep Foundation's sleep quality recommendations: first report. Sleep Health. 2017 Feb;3(1):6-19. doi: 10.1016/j.sleh.2016.11.006. Epub 2016 Dec 23. PMID 28346153
- [Result] Ohayon MM, Paiva T. Global sleep dissatisfaction for the assessment of insomnia severity in the general population of Portugal. Sleep Med. 2005 Sep;6(5):435-41. doi: 10.1016/j.sleep.2005.03.006. PMID 16085459
- [Result] Patel D, Steinberg J, Patel P. Insomnia in the Elderly: A Review. J Clin Sleep Med. 2018 Jun 15;14(6):1017-1024. doi: 10.5664/jcsm.7172. PMID 29852897
- [Result] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Result] Vagharseyyedin SA, Salmabadi M, BahramiTaghanaki H, Riyasi H. The impact of self-administered acupressure on sleep quality and fatigue among patients with migraine: A randomized controlled trial. Complement Ther Clin Pract. 2019 May;35:374-380. doi: 10.1016/j.ctcp.2018.10.011. Epub 2018 Oct 19. PMID 30600173
- [Result] Yin C, Buchheit TE, Park JJ. Acupuncture for chronic pain: an update and critical overview. Curr Opin Anaesthesiol. 2017 Oct;30(5):583-592. doi: 10.1097/ACO.0000000000000501. PMID 28719458
- [Result] Yeung WF, Chung KF, Leung YK, Zhang SP, Law AC. Traditional needle acupuncture treatment for insomnia: a systematic review of randomized controlled trials. Sleep Med. 2009 Aug;10(7):694-704. doi: 10.1016/j.sleep.2008.08.012. Epub 2009 Mar 19. PMID 19303356
- [Result] Yang MH, Lin LC, Wu SC, Chiu JH, Wang PN, Lin JG. Comparison of the efficacy of aroma-acupressure and aromatherapy for the treatment of dementia-associated agitation. BMC Complement Altern Med. 2015 Mar 29;15:93. doi: 10.1186/s12906-015-0612-9. PMID 25880034